CLINICAL TRIAL: NCT03329170
Title: Improved Oral Health in Children with Congenital Heart Disease - an Educational Intervention Trial to Maintain Good Oral Health and Dental Care in Children with Congenital Heart Disease
Brief Title: Improved Oral Health and Dental Care in Children with Congenital Heart Disease
Acronym: ORALPEDHEART
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: My Blomqvist (Other)
Responsible Party: Sponsor-Investigator, My Blomqvist, DDS, Specialist in Paediatric Dentistry, PhD, Helsinki University Central Hospital
Organization: Helsinki University Central Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ORALPEDHEART
Record Dates: First submitted 2017-10-10; First posted 2017-11-01 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Oral Health; Dental Caries
Keywords: Oral health; Dental caries; Heart Defects; Congenital
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- CHD intervention (Experimental): educational intervention using motivational interviewing
  Interventions: Behavioral: educational intervention using motivational interviewing
- CHD control (No Intervention): At 24 and 36 months of age the parents of the child will fill in a questionnaire via internet, designed to assess oral health behaviour. At 36 months of age the child will be offered to participate in a clinical dental examination.
- Healthy control (No Intervention): At 36 months of age the parents of the child will fill in a questionnaire via internet, designed to assess oral health behaviour. At 36 months of age the child will be offered to participate in a clinical dental examination.

INTERVENTIONS:
Behavioral: educational intervention using motivational interviewing — A dental hygienist will offer the families verbal and written information regarding oral health and its importance in children with CHD at the cardiac ward, when child is <12 months. At 6, 12 and 18 months of age, oral health behaviour is assessed via internet, the parents of the child will be sent written information regarding oral health, a tooth brush and a 1000ppm Fluoride tooth paste, after which the dental hygienist will call the parents of the child, to provide additional counselling regarding oral health and its importance in children with CHD. The counselling will be done by motivational interviewing. The themes discussed will be the parents' concerns regarding main points in the written information from the cardiac ward: oral home care, eating habits and dental contact.
  Arms: CHD intervention

SUMMARY:
Background: Congenital heart disease (CHD) is one of the most common congenital anomalies in children. As the risk for endocarditis following bacteraemia is more common during daily oral hygiene routines, such as tooth brushing, than during dental treatment, the maintenance of optimal oral health in children with CHD may be considered of outmost importance. Children with CHD have a higher caries prevalence compared to healthy controls.

Aim: The primary aim of the study is to explore if an educational intervention including information, counselling and support provided at early stage to families affected by major CHD, or CHD combined with a syndrome, can increase the awareness of the importance of maintaining of good oral health, and avoid the development of poor oral health including dental caries, leading to less dental anxiety and a higher oral heath related quality of life. The secondary aim is to elucidate factors associated with the development of poor oral health and/or orofacial dysfunction as well as family attitudes and needs of support.

Hypothesis: Early information, counselling and support will lead to a) increased awareness of the importance to maintaining good oral health, b) prevent the development of poor oral health and dental caries, c) lead to less dental fear, and d) lead to higher oral heath related quality of life.

Study design: Randomized educational intervention trial. Study population: Children born in Finland and under 12 months of age in 1.7.2017-31.12.2021 with, a) major CHD and potentially included in the criteria of endocarditis prophylaxis, or b) with a major CHD combined with a chromosomal syndrome, will be offered to participate in the study. Patients will be recruited until 200 patients are obtained at the Helsinki University Children's Hospital. A control group consisting of approximately 100 healthy children will also be recruited at birth.

Main outcomes: Dental caries, dental anxiety, oral health related quality of life, and awareness of importance to maintain and behaviour to maintain good oral health.

Significance: Better information to patients leads to better possibility to achieve good oral health. Better oral health leads to 1) less dental procedures and thereby less dental anxiety, 2) less dental procedures under general anaesthesia, which may potentially be a risk procedure for the child with CHD, and 3) better oral health related quality of life.

DETAILED DESCRIPTION:
Power analysis:

Children with CHD are at high risk of developing caries (Stecksén-Blicks C et al 2004). In Swedish high-risk areas for developing caries, 12 % of three-year-old children had moderate and severe carious lesions (ICDAS II 3-6) and 11% initial carious lesions (ICDAS II 1-2) (Anderson et al 2016). Based on the assumption that 10% in the intervention group and 30% in the control group will develop caries (ICDAS II 1-6), p<0.05 and power 0.80, a sample size of at least 65 individuals in each age group is required. 1.7.2017-31.12.2021 198 Finnish speaking families will be offered to participate in the study. To secure an even distribution block randomization will be used. The patients will be randomized into blocks of 4 and 8, with the help of www.randomization.com (Pandis et al 2011).

ELIGIBILITY:
Inclusion criteria:

* Age < 12 months and prostethic cardiac valve or patient likely to undergo valve surgery using foreign material including homograft (potentially included in the criteria of endocarditis prophylaxis)
* Age < 12 months and unrepaired cyanotic CHD including palliative shunts and conduits
* Age < 12 months and repaired CHD with residual defects at the site or adjacent to the site of the prosthetic patch or device which inhibits endothelialization
* Age < 12 months and cardiac transplantation recipient or listed for transplantation (potentially included in the criteria of endocarditis prophylaxis)
* Age < 12 months and cardiomyopathy (potential cardiac transplantation recipient)
* Age < 12 months and chromosomal abnormality or syndrome and any invasive intevention (surgery or cath) for CHD or likely to require invasive intervention for CHD

Exclusion criteria:

* Neither parent amenable to comprehend intervention instructions provided in Finnish
* Child in out-of-home care (eg foster care)

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Caries | 36 months of age
  During a clinical dental examination, caries will be registered clinically according to the ICDAS II (Pitts et al 2013, Shoaib et al 2009). The caries lesions on a tooth surface are graded as "initial" (ICDAS 1-2), "moderate" (ICDAS 3-4) and "extensive" (ICDAS 5-6). The indexes dmfs (decayed, missing or filled surfaces) and dmft (decayed, missing or filled surfaces) will be calculated separately for ICDAS 1-2, ICDAS 3-6 and ICDAS 1-6. The range for dmfs is 0-88 and dmft is 0-20, with 0 indicating no caries, and an increasing number indicating more carious lesions.
Dental plaque | 36 months of age
  During a clinical dental examination, visible plaque will be registered on the labial surfaces of the maxillary incisors (y/n) as a risk indicator for developing caries (Alaluusua and Malmivirta 1994).
Awareness of the importance to maintain good oral heath | Intervention group at 24 and 36 months of age; CHD control group at 24 and 36 months of age; healthy control group at 24 and 36 months of age.
  Awareness of the importance to maintain good oral health will be measured with a questionnaire designed to assess adherence to the recommendations in the written information regarding oral health care provided at baseline in the intervention group. The questionnaire includes three domains: tooth brushing, sugar intake, and dental contact. Tooth brushing includes 6 questions (morning, night, parent brushing, problems with brushing, continue brushing though problems, fluoride tooth paste), sugar intake includes 5 questions (frequency of eating, sugary drink, eating during night, sugary food, medicine taken with sugar), and the dental contact includes one question (dental visit). Every answer not in accordance to the recommendations given, is scored with 1 point, giving a range in tooth brushing 0-6, sugar intake 0-5, and dental contact 0-1, with an increasing value indicating less awareness of the importance to maintain good oral health.

SECONDARY OUTCOMES:
Developmental defects of the enamel | 36 months of age
  During a clinical dental examination, developmental defects of the enamel will be registered clinically according to the modified DDE index (Fédération Dentaire Internationale 1992). The Modified Developmental Defects of Enamel Index (Modified DDE Index) is used to diagnose and classify changes in the enamel of the deciduous teeth studied. Three surfaces are examined: buccal, occlusal/incisal and lingual/palatal of all deciduous teeth. The enamel defects are assessed according to three clinical aspects: hypoplasia of the enamel (3 types), diffuse opacities (4 types) and demarcated opacities (2 types). The extent of the affected area is registered in three grades. Number of teeth affected (n) in one patient is then counted.
Orofacial dysfunction | 36 months of age
  Orofacial dysfunction, such as difficulties to speak, chew, or swallow, is screened for using The Nordic Orofacial Test - Screening (NOT-S). NOT-S consist of a structured interview and a clinical examination where an illustrated manual is to be used. The NOT-S interview contains six domains: sensory function, breathing, habits, chewing and swallowing, drooling, and dryness of the mouth (I-VI). NOT-S examination contains six domains representing: face at rest, and tasks regarding nose breathing, facial expression, masticatory muscle and jaw function, oral motor function, and speech (1-6). One or more "yes" for impairment in a domain results in one point (maximum NOT-S score 12 points). Normal data for children typically vary between 0 and 4, with a higher value indicating more orofacial dysfunction. The NOT-S test situation will be video recorded, and the analysis will be done by a blinded speech therapist.
Dental fear | 36 months of age
  Dental anxiety in the child will be measured by Children's' Fear Survey Schedule-Dental subscale (CFFS-DS). The CFSS-DS questionnaire covers different aspects of dental and medical treatment situations and consists of 15 items. The response to each question is a score from 1 (not afraid) to 5 (very afraid), with a total score varying between 15 and 75. Children with a CFSS-DS score of more than or equal to 38 are defined as dentally anxious.
  Parental dental anxiety will be measured by the Modified Dental Anxiety Scale (MDAS). MDAS comprises five multiple-choice questions addressing the individual's reactions and expectations of going to and being treated by a dentist. Each question consists of 5 response alternatives ranging from 1 (no anxiety) to 5 (extreme anxiety) with a total score varying between 5 and 25. A MDAS score of 19-25 indicates high dental anxiety.
Oral health related quality of life (OHRQoL) | 36 months of age
  The Parental- Caregivers Perception Questionnaire (P-CPQ) is used to measure he child's oral health related quality of life (OHRQoL), and has the following domains: Oral symptoms (7 items), Functional limitations (7 items), Emotional well-being (9 items) and Social well- being (10 items). Each question has 5 response options (0-4). Total score range 0-124. Scores for domains can be computed separately. A higher score indicates a greater negative OHRQoL of the child.
  The Family Impact Scale (FIS) is used to measure the effect of the child's oral health on the family. The FIS consists 12 items divided into three subscales: parental/family activity (5 items), parental emotions (3 items) and family conflict (4 items), and 2 global questions concerning oral health and general well-being. Each question has 5 response options (0-4). Total FIS score range 0-56, where a higher score denotes greater impact of a child's oral condition on family QoL.

CONTACTS AND LOCATIONS:
Overall Officials: My Blomqvist, PhD, Principal Investigator — Department of Oral and Maxillofacial Diseases, Helsinki University Central Hospital.
Locations (1):
- Department of Pediatrics, Children´s Hospital, Helsinki University Central Hospital., Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No